CLINICAL TRIAL: NCT00002916
Title: A Phase II Trial in Patients With Early Cervical Cancer to Study The Safety and The Immunological Effects of Vaccination With TA-HPV, A Live Recombinant Vaccinia Virus Expressing The Human Papilloma Virus 16 and 18 E6 and E7 Proteins
Brief Title: Surgery and Vaccine Therapy in Treating Patients With Early Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-13961; EORTC-13961
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Cervical Cancer
Keywords: stage IB cervical cancer; stage IIA cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — oncogene protein E7, Human papillomavirus type 16; E6 protein, Human papillomavirus type 16; Chemotherapy, Adjuvant; Surgical Procedures, Operative; Radiotherapy

INTERVENTIONS:
Biological: human papillomavirus 16 E7 peptide
Biological: synthetic human papillomavirus 16 E6 peptide
Procedure: adjuvant therapy
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Vaccines made from human papillomavirus may make the body build an immune response to and kill cervical cancer cells. Combining vaccine therapy with surgery may be a more effective treatment for cervical cancer.

PURPOSE: This phase II trial is studying how well giving vaccine therapy together with surgery works in treating patients with early cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the systemic immunological response to the human papilloma virus vaccine (TA-HPV) expressing the proteins 16, 18, E6 and E7 examining the cytolytic T cell and the antibody responses in cervical cancer patients.
* Investigate further the safety and toxic effects of TA-HPV in these patients.
* Assess the proliferative capacity of T cells to the E6 and E7 proteins.
* Observe any influence of vaccination with TA-HPV on the disease free interval or patterns of recurrence in these patients.

OUTLINE: This is an open-label, nonrandomized study.

Patients receive 2 vaccinations of the human papilloma virus with proteins 16, 18, E6 and E7 at least 4 weeks apart, with the first vaccination at least 2 weeks before surgery and the second 8 weeks after the first one, unless unacceptable toxicity occurs. Patients who require radiotherapy following surgery receive their second vaccination 4-8 weeks after the first vaccination.

Twenty-eight patients are entered initially; if at least 2 patients show an immunologic response, 16 additional patients are entered.

Patients are followed every 3 months for 2 years, then every 6 months for 3 years, then annually.

PROJECTED ACCRUAL: 44 patients will be entered over 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven untreated stage Ib or IIa cervical carcinoma, squamous or adenocarcinoma suitable for surgical excision

  * No CNS metastases
* Circulating CD4+ lymphocyte count at least 400
* Proven absence of hepatitis B and C antibodies
* Previous exposure to vaccinia from smallpox vaccination, as well as no previous exposure, is allowed
* Reaction to 2 or more antigens on Pasteur Merieux CMI test required
* Ability to collaborate planned follow-up required

PATIENT CHARACTERISTICS:

Age:

* 19 and over

Performance status:

* WHO/ECOG no greater than 2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC greater than 3,000 (3,000 x 10 to the ninth/L)
* Platelet count greater than 120,000 (120 x 10 to the ninth/L)
* No bleeding disorder

Hepatic:

* Bilirubin less than 1.5 times normal
* AST and ALT less than 1.5 times normal
* Prothrombin or partial thromboplastin time no greater than 2 times normal

Renal:

* Creatinine less than 1.3 mg/dL (120 micromoles/L)

Other:

* No ongoing infection
* No HIV antibody
* No serious medical or psychiatric illness
* No second malignancy within 5 years except for curatively treated basal cell skin cancer which required surgery, hormone therapy, immunotherapy or chemotherapy
* Not pregnant or nursing
* Adequate contraception required
* Patient or her household contacts must not have any of the following:

  * Chronic steroid therapy
  * Renal or other allograft
  * Known immunodeficiency
  * Eczema
  * Children under 5 years old

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 1996-11

PRIMARY OUTCOMES:
Immunological response to HPV
Toxicity and safety of TA-HPV

SECONDARY OUTCOMES:
Proliferative capacity of T-cells to the E6 and E7 proteins
Influence of vaccination with TA-HPV on the disease free interval or patterns of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Elaine M. Rankin, MD, Study Chair — Ninewells Hospital
Locations (10):
- Innsbruck Universitaetsklinik, Innsbruck, Austria
- Institut Curie - Section Medicale, Paris, France
- Germany (2):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - I. Frauenklinik und Hebammenschule der Ludwig-Maximillians Universitaet Muenchen, Munich
- Nijmegen Cancer Center at Radboud University Medical Center, Nijmegen, Netherlands
- Norwegian Radium Hospital, Oslo, Norway
- University Hospital of Linkoping, Linköping, Sweden
- United Kingdom (3):
  - St. Mary's Hospital, Manchester, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Velindre Cancer Center at Velinde Hospital, Cardiff, Wales